CLINICAL TRIAL: NCT00493298
Title: TOP: TYSABRI Observational Program
Brief Title: Tysabri Observational Program
Acronym: TOP
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: IMA-06-02
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: disease progression; Multiple Sclerosis; disease activity; Tysabri; natalizumab; long-term safety
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Disease Progression; Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tysabri: According to the local prescribing information
  Interventions: Drug: Tysabri

INTERVENTIONS:
Drug: Tysabri — According to the local prescribing information
  Other Names: BG00002; natalizumab

SUMMARY:
The primary objective of this study is to assess the long-term safety and impact on disease activity and progression of Tysabri in participants with relapsing remitting multiple sclerosis (RRMS) in a clinical practice setting.

DETAILED DESCRIPTION:
TOP is an epidemiological observational study of participants receiving natalizumab, with each participant to be followed for up to 15 years. This study is designed to address the long-term safety profile and the long-term impact on disease activity and progression of Tysabri with marketed use, and the impact of treatment on disability in particular by comparing the results with prospectively determined controls from established databases.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of Relapsing Remitting Multiple Sclerosis
* The decision to treat with Tysabri must precede enrollment
* Patient must be a new Tysabri user, and must not have had more than 3 Tysabri infusions prior to enrollment
* Must have had at least one relapse in the previous year, and must satisfy locally approved therapeutic indications for Tysabri

Key Exclusion Criteria:

* History of Progressive Multifocal Leukoencephalopathy or other opportunistic infections, or an increased risk of opportunistic infections
* History of positive anti-Tysabri antibodies
* Concomitant Immunomodulatory or immunosuppressive therapy during therapy with Tysabri
* Patient immunocompromised at the time of enrollment
* Known active malignancy
* Women must not be breast feeding or pregnant, or planning to become pregnant (must use birth control unless surgically sterile)

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with RRMS who are therapy-naïve to Tysabri and who meet the criteria defined in the indication statement for prescription in the respective country.
Sampling Method: Non-Probability Sample
Enrollment: 6620 (Actual)
Dates: Start 2007-06-29 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious Adverse Events (SAE) | Up to 15 years

SECONDARY OUTCOMES:
Annualized Relapse Rate (ARR) | Yearly for up to 15 years
  A clinical relapse is defined as new or recurrent neurological symptoms, not associated with fever, lasting for at least 24 hours, and followed by a period of 30 days of stability or improvement. New or recurrent neurological symptoms that occur less than 30 days following the onset of a protocol-defined relapse should be considered part of the same relapse.
Distribution of the Total Number of Relapses | Yearly for up to 15 years
Time to First Relapse | Yearly for up to 15 years
Percentage of Participants with Relapse | Yearly for up to 15 years
Percentage of Participants with Disability Progression | Yearly for up to 15 years
  Disability progression is defined as at least a 1.0 point increase on the Expanded Disability Status Scale (EDSS) from Baseline that is sustained over 6 months. The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist.
Percentage of Participants that reach Expanded Disability Status Score (EDSS) Milestones Indicating Increasing Disability | Yearly for up to 15 years
  The percentage of participants that reach EDSS milestones such as 4.0, 6.0, and 7.0 sustained after 6 months. The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist.
Percentage of Participants whose EDSS Worsened, Stabilized or Improved and Sustained over 6 Months | Yearly for up to 15 years
Evaluation of Baseline Disease Characteristics as Prognostic Indicators for Disease Activity and Disability Progression Over Time | Yearly for up to 15 years
  Baseline disease characteristics evaluated will include: EDSS; Disease duration at baseline; Number of relapses during 1 and 2 years before baseline; Previous use of disease modifying therapy; Age, gender.
Evaluation of Short-Term (1 year) Disease Outcomes as Prognostic Indicators for Disease Activity and Disability Progression Over Time | Yearly for up to 15 years
  Short term outcomes evaluated will include: EDSS progression during first 12 months; Occurrence of relapses during first 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (355):
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Córdoba
  - Research site, Santa Fe
- Australia (14):
  - Research site, Camperdown, New South Wales
  - Research site, Liverpool, New South Wales
  - Research site, New Lambton Heights, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Auchenflower, Queensland
  - Research site, Gold Coast, Queensland
  - Research site, Adelaide, South Australia
  - Research Site, North Adelaide, South Australia
  - Research site, Box Hill, Victoria
  - Research site, Fitzroy, Victoria
  - Research site, Heidelberg, Victoria
  - Research Site, Melbourne, Victoria
  - Research site, Parkville, Victoria
  - Research site, Nedlands, Western Australia
- Belgium (29):
  - Research site, Aalst
  - Research site, Anderlecht
  - Research site, Antwerp
  - Research site, Bocholt
  - Research site, Brasschaat
  - Research site, Bruges
  - Research site, Brussels
  - Research site, Charleroi
  - Research Site, Charleroi
  - Research site, Edegem
  - Research site, Fraiture
  - Research site, Genk
  - Research site, Ghent
  - Research site, Hasselt
  - Research site, Jette
  - Research site, Kortrijk
  - Research site, La Louvière
  - Research site, Leuven
  - Research site, Libramont
  - Research site, Liège
  - Research site, Malmedy
  - Research site, Melsbroek
  - Research site, Ostend
  - Research site, Ottignies
  - Research Site, Overpelt
  - Research site, Sijsele
  - Research site, Tournai
  - Research site, Wilrijk
  - Research site, Woluwe-Saint-Lambert
- Brazil (4):
  - Research Site, Belo Horizonte
  - Research Site, Botucatu
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (17):
  - Research site, Edmonton, Alberta
  - Research site, Burnaby, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research site, Winnipeg, Manitoba
  - Research site, Saint John, New Brunswick
  - Research site, Halifax, Nova Scotia
  - Research site, Bracebridge, Ontario
  - Research site, Guelph, Ontario
  - Research site, Hamilton, Ontario
  - Research site, London, Ontario
  - Research site, Milton, Ontario
  - Research site, Thunder Bay, Ontario
  - Research site, Toronto, Ontario
  - Research site, Gatineau, Quebec
  - Research site, Greenfield Park, Quebec
  - Research site, Montreal, Quebec
  - Research site, Regina, Saskatchewan
- Czechia (12):
  - Research site, Brno
  - Research site, České Budějovice
  - Research site, Hradec Kralové
  - Research site, Jihlava
  - Research site, Olomouc
  - Research site, Ostrava
  - Research site, Pardubice
  - Research site, Pilsen
  - Research site, Prague
  - Research site, Teplice
  - Research Site, Teplice
  - Research site, Zlín
- Finland (7):
  - Research site, Helsinki
  - Research site, Jyväskylä
  - Research site, Kuopio
  - Research site, Pori
  - Research site, Seinäjoki
  - Research site, Tampere
  - Research site, Turku
- France (60):
  - Research site, Agen
  - Research site, Aix-en-Provence
  - Research site, Alençon
  - Research site, Angoulême
  - Research site ,1 Allée du Château- Dr Wagner, Ars-Laquenexy
  - Research site, Auxerre
  - Research site, Avranches
  - Research site, Bayonne
  - Research site, Beauvais
  - Research site, Belfort
  - Research site, Beuvry
  - Research site, Béthune
  - Research site, Boulogne-sur-Mer
  - Research site, Calais
  - Research site, Castelnau-le-Lez
  - Research site, Castres
  - Research site, Chambéry
  - Research site, Colmar
  - Research site, Compiègne
  - Research site, Dieppe
  - Research site, Dreux
  - Research site, Dunkirk
  - Research site, Épinal
  - Research site, Évreux
  - Research site, Haguenau
  - Research site, La Rochelle
  - Research site 177, rue de Versailles- Dr Servan, Le Chesnay
  - Research site, Le Chesnay
  - Research site, Le Coudray
  - Research site, Le Havre
  - Research site, Le Mans
  - Research site, Lille
  - Research site, Lisieux
  - Research site, Lomme
  - Research site, Mantes-la-Jolie
  - Research site, Maubeuge
  - Research site, Metz
  - Research site, Metz-Tessy
  - Research site, Mont-de-Marsan
  - Research site, Montauban
  - Research site, Montluçon
  - Research site, Montpellier
  - Research site, Mulhouse
  - Research site, Nice
  - Research site, Paris
  - Research site, Pau
  - Research site, Quimper
  - Research site, Reims
  - Research site, Saint-Aubin-sur-Scie
  - Research site, Sarreguemines
  - Research site, Saumur
  - Research site, St-Malo
  - Research site, Talant
  - Research site, Tarbes
  - Research site, Tourcoing
  - Research site, Trappes
  - Research site, Trélazé
  - Research site, Valenciennes
  - Research site, Vesoul
  - Research site, Vichy
- Germany (100):
  - Research site, Abensberg
  - Research site, Andernach
  - Research Site, Arnsdorf
  - Research site, Asperg
  - Research site, Augsburg
  - Research site, Bad Hersfeld
  - Research site, Bad Honnef
  - Research Site, Bad Kissingen
  - Research site, Bad Mergentheim
  - Research site, Bad Reichenhall
  - Research site, Bamberg
  - Research site, Berlin
  - Research site, Bielefeld
  - Research site, Bochum
  - Research site, Bogen
  - Research site, Bonn
  - Research site, Bruchsal
  - Research site, Buchholz
  - Research site, Celle
  - Research site, Chemnitz
  - Research site, Cologne
  - Research site, Dillingen
  - Research site, Dresden
  - Research site, Duisburg
  - Research site, Düren
  - Research site, Düsseldorf
  - Research site, Eisenach
  - Research site, Emden
  - Research site, Emmendingen
  - Research site, Erbach im Odenwald
  - Research site, Erlangen
  - Research site, Essen
  - Research site, Falkenstein
  - Research site, Frankfurt
  - Research site, Freiburg im Breisgau
  - Research site, Görlitz
  - Research site, Göttingen
  - Research site, Greifswald
  - Research site, Halle
  - Research site, Hamburg
  - Research site, Heidelberg
  - Research site, Herford
  - Research site, Itzehoe
  - Research site, Jena
  - Research site, Kaiserslautern
  - Research site, Kaltenkirchen
  - Research site, Kandel
  - Research site, Kassel
  - Research site, Kastellaun
  - Research site, Kirchberg
  - Research site, Kirchheim unter Teck
  - Research Site, Kreuzau
  - Research site, Ladenburg
  - Research site, Leipzig
  - Research site, Lengerich
  - Research site, Ludwigshafen
  - Research site, Lüdenscheid
  - Research site, Lüneburg
  - Research site, Magdeburg
  - Research site, Mannheim
  - Research site, Marburg
  - Research site, München
  - Research site, Münster
  - Research site, Neuburg am Inn
  - Research site, Neukirchen-Vluyn
  - Research site, Neuruppin
  - Research site, Nuremberg
  - Research site, Oldenburg
  - Research site, Olpe
  - Research site, Osnabrück
  - Research site, Paderborn
  - Research site, Potsdam
  - Research site, Regensburg
  - Research site, Remscheid
  - Research site, Rüdersdorf
  - Research Site, Rülzheim
  - Research site, Schlüchtern
  - Research site, Schorndorf
  - Research site, Schwaebisch
  - Research site, Siegen
  - Research site, Sinsheim
  - Research site, Stade
  - Research site, Stadtroda
  - Research site, Stuttgart
  - Research site, Tegel
  - Research site, Teupitz
  - Research site, Trier
  - Research site, Troisdorf
  - Research site, Ulm
  - Research site, Unterhaching
  - Research site, Wasserburg
  - Research site, Weimar
  - Research site, Weinheim
  - Research site, Wermsdorf
  - Research site, Wernigerode
  - Research site, Wiesbaden
  - Research site, Wolfenbüttel
  - Research site, Wolfratshausen
  - Research site, Würzburg
  - Research site, Zwickau
- Greece (6):
  - Research site, Heraklion, Crete
  - Research Site, Alexandroupoli
  - Research site, Athens
  - Research site, Ioannina
  - Research site, Pátrai
  - Research site, Thessaloniki
- Italy (14):
  - Research site, Bari
  - Research site, Bergamo
  - Research site, Cagliari
  - Research site, Cefalù
  - Research site, Chieti
  - Research site, Cuneo
  - Research site, Fidenza
  - Research site, Florence
  - Research site, Foggia
  - Research site, Gallarate
  - Research site, Milan
  - Research site, Napoli
  - Research site, Orbassano
  - Research site, Roma
- Mexico (10):
  - Research site, Zapopan, Jalisco
  - Research site, Monterrey, Nuevo León
  - Research site, Aguascalientes
  - Research site, Estado de México
  - Research Site, León
  - Research site, Mexico City
  - Research Site, Mexico City
  - Research site, Puebla City
  - Research Site, Puebla City
  - Research Site, San Luis Potosí City
- Netherlands (24):
  - Research site, 's-Hertogenbosch
  - Research Site, Almelo
  - Research site, Blaricum
  - Research site, Breda
  - Research site, Eindhoven
  - Research site, Geldrop
  - Research site, Gouda
  - Research site, Heerenveen
  - Research site, Heerlen
  - Research site, Helmond
  - Research site, Hengelo
  - Research site, Hoorn
  - Research site, Leeuwarden
  - Research Site, Meppel
  - Research site, Nieuwegein
  - Research site, Nijmegen
  - Research site, Roermond
  - Research site, Rotterdam
  - Research site, Sittard-Geleen
  - Research site, The Hague
  - Research site, Tilburg
  - Research site, Venray
  - Research site, Woerden
  - Research Site, Zwolle
- Norway (17):
  - Research site, Bergen
  - Research site, Bodø
  - Research site, Drammen
  - Research Site, Fredrikstad
  - Research site, Førde
  - Research site, Haugesund
  - Research site, Lillehammer
  - Research site, Lørenskog
  - Research site, Molde
  - Research site, Namsos
  - Research site, Oslo
  - Research Site, Oslo
  - Research Site, Skien
  - Research site, Stavanger
  - Research Site, Tromsø
  - Research site, Trondheim
  - Research site, Tønsberg
- Portugal (7):
  - Research site, Aveiro
  - Research site, Beja
  - Research site, Evora
  - Research site, Funchal
  - Research site, Lisbon
  - Research site, Porto
  - Research site, Setúbal
- Slovakia (5):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research site, Bratislava
  - Research site, Košice
  - Research site, Nitra
- Spain (11):
  - Research site, Ávila
  - Research site, Badalona
  - Research site, Barcelona
  - Research site, Donostia / San Sebastian
  - Research site, Girona
  - Research site, Langreo
  - Research site, Logroño
  - Research site, Palma de Mallorca
  - Research site, Ponferrada
  - Research site, Tarragona
  - Research site, Vitoria-Gasteiz
- United Kingdom (14):
  - Research site, Edgbaston, Birmingham
  - Research site, Canterbury, Kent
  - Research site, Hammersmith, London
  - Research site, Salford, Manchester
  - Research site, Belfast
  - Research site, Brighton
  - Research site, Bristol
  - Research site, Coventry
  - Research site, Exeter
  - Research site, Liverpool
  - Research site, Middlesbrough
  - Research site, Newcastle upon Tyne
  - Research site, Nottingham
  - Research site, Stoke-on-Trent

REFERENCES:
- [Derived] Butzkueven H, Kappos L, Spelman T, Trojano M, Wiendl H, Su R, Liao S, Hyde R, Licata S, Ho PR, Campbell N. No evidence for loss of natalizumab effectiveness with every-6-week dosing: a propensity score-matched comparison with every-4-week dosing in patients enrolled in the Tysabri Observational Program (TOP). Ther Adv Neurol Disord. 2021 Sep 27;14:17562864211042458. doi: 10.1177/17562864211042458. eCollection 2021. PMID 34603507
- [Derived] Butzkueven H, Kappos L, Wiendl H, Trojano M, Spelman T, Chang I, Kasliwal R, Jaitly S, Campbell N, Ho PR, Licata S; Tysabri Observational Program (TOP) Investigators. Long-term safety and effectiveness of natalizumab treatment in clinical practice: 10 years of real-world data from the Tysabri Observational Program (TOP). J Neurol Neurosurg Psychiatry. 2020 Jun;91(6):660-668. doi: 10.1136/jnnp-2019-322326. Epub 2020 Mar 31. PMID 32234967
- [Derived] Butzkueven H, Kappos L, Pellegrini F, Trojano M, Wiendl H, Patel RN, Zhang A, Hotermans C, Belachew S; TYSABRI Observational Program (TOP) Investigators. Efficacy and safety of natalizumab in multiple sclerosis: interim observational programme results. J Neurol Neurosurg Psychiatry. 2014 Nov;85(11):1190-7. doi: 10.1136/jnnp-2013-306936. Epub 2014 Feb 14. PMID 24532785